CLINICAL TRIAL: NCT00601601
Title: Genomics Approach to Id Novel Targets & Markers for Early Detection And Intervention In Cancer (Cervical)
Brief Title: Identifying Biomarkers for Early Detection of Cancer in Patients With Cervical Dysplasia or Carcinoma in Situ of the Cervix
Status: Completed | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000581302; R01CA103830 (NIH); BCCR-H04-60112; BCCR-RO4-0112
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: stage 0 cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tissue from patients with abnormal cells may help doctors identify biomarkers related to cancer.

PURPOSE: This clinical trial is identifying biomarkers for early detection of cancer in women with cervical dysplasia or carcinoma in situ of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify and catalogue genetic alterations and protein changes associated with developmental stages of cervical cancer.
* To identify a ranked list of candidate genes that drive the transformation of premalignant lesions to tumors for further study and validation as molecular targets for novel early detection and treatment design.

Secondary

* To complete genome scans at high density and analysis of gene and protein expression to identify recurrent genetic and protein changes in cancer.
* To confirm changes clustered to specific chromosomal regions which harbor tumor suppressors or oncogenes.

OUTLINE: Patients undergo biopsy of cervical tissue followed by loop electrocautery excision procedure (LEEP) (removing all of the tissue surrounding and under the area biopsied). RNA, DNA, and protein is extracted from the cells to provide material for the construction of libraries for Serial Analysis of Gene Expression (SAGE analysis); for hybridization against Bacterial Artificial Chromosome Comparative Genome Hybridization arrays (BAC CGH arrays); and for analysis using protein chip arrays and proteomics. Resulting data from coded samples provide gene expression and protein profiles. The coded molecular datasets are linked, analyzed, and compared using a variety of statistical software to identify putative genes, gene alterations, and proteins of interest. Some samples may be banked for future studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed premalignant lesion, dysplasia, or carcinoma in situ of the cervix
* Clinically documented disease
* Attending Vancouver General Hospital and referred to colposcopy for loop electrocautery excision procedure (LEEP)

PATIENT CHARACTERISTICS:

* Not pregnant
* No lack of informed consent due to language difficulty, physical and mental condition

PRIOR CONCURRENT THERAPY:

* No prior operation for removal of the cervix
* Concurrent therapy allowed

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending Vancouver General Hospital and referred to colposcopy for loop electrocautery excision procedure (LEEP).
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2004-12; Primary Completion 2009-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Identify and catalogue genetic alterations and protein changes associated with developmental stages of cervical cancer | Done at the completion of the study.
Identify a ranked list of candidate genes that drive the transformation of premalignant lesions to tumors for further study and validation as molecular targets for novel early detection and treatment design | Done at the completion of the study.
Completion of genome scans at high density and analysis of gene and protein expressions to identify recurrent genetic and protein changes in cancer | Done at the completion of the study.
Changes clustered to specific chromosomal regions which harbor tumor suppressors or oncogenes | Done at the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lam, Study Chair — British Columbia Cancer Agency